CLINICAL TRIAL: NCT02813330
Title: Subcutaneous Sterile Water Injection for Relief of Low Back Pain During Normal Labor: Randomized Controlled Study
Brief Title: Subcutaneous Sterile Water Injection for Relief of Low Back Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Howieda Fouly, PhD, Lecturer of Obstetric & gynecological nursing, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Women Health Hospital
Record Dates: First submitted 2016-06-18; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Low Back Pain
Keywords: Women; severe; low back ache; labor
MeSH Terms: conditions — Low Back Pain; Lymphoma, Follicular | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sterile Water injection (Experimental): Subcutenous injection at low back portion during labor pain
  Interventions: Other: Subcutaneous sterile water injection; Other: saline injection
- saline injection (Experimental): Subcutenous injection at low back portion during labor pain
  Interventions: Other: Subcutaneous sterile water injection; Other: saline injection

INTERVENTIONS:
Other: Subcutaneous sterile water injection — sterile water injection in two points of low back pain
  Other Names: sterile water injection
Other: saline injection — Saline injection in two points of low back pain
  Other Names: Natural pain relief

SUMMARY:
To compare the effect of subcutenous sterile water injection technique with the subcutaneous saline injection technique in the degree and duration of low back pain-relieving during childbirth

DETAILED DESCRIPTION:
Study sample:

The convenience sample will be recruited randomly on the basic of odd number will have saline injection and even number will be given a placebo (Sterile water injection)

Setting:

Labor ward in Women's health center at Assiut university hospital

Study design:

Experimental Randomized control study

Sample size:

The sample size was calculated using the formula N= (Zα+Zβ)2 x 2p(1-p)÷d2 ,taking the level of significance as 5%, Zα=1.96 and power of the test as 80%, Zβ=0.84. p=0.113. A sample size of 165 in each group was calculated. Total of 330 women will be studied (165 in each arm) Inclusion criteria

* In labour (spontaneous or induced
* During first stageof labour
* Primary and multiparous women
* A term singleton pregnancy (between 37 + 0 and 41 weeks)
* Have a fetus in a cephalic presentation
* Experience back pain assessed by visual analogue scale VAS and Face pain analogue ( Warden V, Hurley AC, Volicer L.2003)
* Provide informed consent.

Exclusion criteria

* Multiple pregnancy
* Malpresentation (breech, transverse, shoulder)
* Previous CS
* Infection or inflammation at the injection sites or complications that could cause bleeding at injection site eg. Thrombocytopenia.

Study Tools:

1. Personal data questionnaire
2. Visual Analogue Scale and Face analogue scale
3. Satisfaction scale

ELIGIBILITY:
Inclusion Criteria:

* In labour (spontaneous or induced record
* During first stage of labour
* Primary and multiparous women
* A term singleton pregnancy (between 37 + 0 and 41 weeks)
* Have a fetus in a cephalic presentation
* Experience back pain assessed by visual analogue scale VAS and Face pain analogue
* Provide informed consent.

Exclusion Criteria:

* Women with chronic disease
* Medical condition associated with pregnancy ( Pre-eclampsia- Eclampsia- Diabetic pregnancy.... etc)
* Complicated labor process ( obstructed, preterm labor, twins)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Pain relief | two hours for each client
  the investigator spend two hours with each client to measure the effect of pain relief
Women's Saisfaction | each 15 min until 120 min
  measuring pain relief within different minutes

IPD SHARING:
Plan to Share IPD: Yes
Protocol or seminar discussion